CLINICAL TRIAL: NCT00105417
Title: A Phase I, Randomized, Placebo-Controlled, Double-Blind Study Evaluating the Safety of Subcutaneous Single Dose Interleukin-7 in HIV-1-Infected Subjects Who Are Receiving Antiretroviral Treatment (A5214)
Brief Title: Interluekin-7 to Treat HIV-Infected People Receiving Antiretroviral Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050112; 05-I-0112
Record Dates: First submitted 2005-03-11; First posted 2005-03-14 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-05

CONDITIONS: HIV Infections; HIV
Keywords: Immune Reconstitution; Thymus; Cytokines; HIV
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-7

INTERVENTIONS:
Drug: IL-7

SUMMARY:
This study will evaluate whether interleukin-7 (IL-7) a drug similar to the natural IL-7 protein produced by the body, is safe to use in people infected with HIV. IL-7 is important in immune system function. In humans, it can extend the life of immune cells called T-cells and increase their function and maturation; in mice, it can speed up immune system recovery following chemotherapy of transplantation; and in monkeys, it can make T-cells increase in numbers. If this study shows that IL-7 is safe, other trials will determine if it can improve the numbers or function of T-cells in HIV-infected people.

Patients 18 years of age and older with HIV infection who have been taking anti-HIV medications for at least 12 months, whose CD4 counts are at least 100 cells/microliter, and whose viral load is no more than 50,000 copies/milliliter may be eligible for this study. Candidates are screened with a physical examination, blood and urine tests, including a blood test for HLA type (a genetic test of markers of the immune system), chest x-ray, electrocardiogram, and ultrasound of the spleen.

Participants undergo the following tests and procedures during 9 visits, as follows:

Pre-entry visit

* Brief physical examination, including examination of lymph nodes and spleen.
* Medical history, including questions about current and past medications.
* Urine pregnancy test for women who are able to become pregnant.
* Blood draw for viral load, immune responses, and other routine safety tests.

Entry visit

* Complete physical examination, including examination of lymph nodes and spleen.
* Routine urine test and urine pregnancy test for women who are able to become pregnant.
* Blood draw for viral load, immune responses, and other routine safety tests.
* IL-7 dosing. Participants are randomly assigned to receive one of five doses of IL-7 (3, 10, 30, 60 or 100 micrograms per kilogram of body weight) or placebo (a salt solution that does not contain IL-7). The dose may be given in one or more injections, with higher doses possibly requiring as many as seven or eight injections. The injections are given subcutaneously (under the skin), usually in the arm or leg. After the injection, patients are monitored closely for 12 hours for skin or allergic reactions. Blood is drawn before the injection and again at 0.5, 1, 1.5, 2, 2.5, 4, 8 and 12 hours after the injection to check blood levels of the study medication.

Follow-up visits

Patients come to the clinic 7 times during follow-up-every day for the first 4 days after the injection, then at 14 days, 4 weeks, and 8 weeks after the injection. At most study visits, patients have the following procedures:

* Brief physical examination, including examination of lymph nodes and spleen.
* Routine urine test and urine pregnancy test for women who are able to become pregnant.
* Blood draw for viral load, immune responses, and other routine safety tests.
* Blood test to measure the amount of study medication in the blood 1, 2, and 3 days after the injection
* Electrocardiogram 1 day after the injection

DETAILED DESCRIPTION:
Interleukin 7 is an essential cytokine for the thymic development and the post-thymic survival, expansion and maturation of the T lymphocytes in humans. Therapeutic use of IL7 in mouse models has shown enhancement of immune reconstitution after chemotherapy or bone marrow transplantation. The rationale for using IL-7 as immunotherapy in HIV infection would be to support the expansion, survival and functional properties of T lymphocytes and enhance immune reconstitution. More specifically, IL7 may provide the means to support CD4 expansions in patients with good viral suppression but persistent low CD4 counts (immunologic non-responders) or in patients who have no available antiretroviral options. Finally, given the role of IL7 in T cell memory maturation and survival, IL-7 may be a promising vaccine adjuvant.

Studies of rhIL7 in non-human primates have shown that T cell proliferation and expansion can be achieved at doses that are well tolerated without significant toxicity. A safety study in cancer patients is currently ongoing at the NCI. A5214 (Pleiades) will be the first study of rhIL7 to evaluate the safety of a single subcutaneous injection in HIV infected adults. Eligible subjects (CD4 greater than 100 cells/micro l and VL less than 50,000 copies/ml, on antiretroviral therapy for at least one year) will be stratified by viral load (less than 50 or 50-50,000 copies/ml) and will be randomized 3:1 to receive rhIL7 or placebo.

Pleiades is a phase I, double-blind trial that will test the safety of a single subcutaneous injection of IL-7 at 5 different doses (3, 10, 30, 60 and 100 micro g/kg) tested sequentially. Four subjects will enroll in each dose level and dose escalation will occur only after all subjects complete four weeks without evidence of dose-limiting toxicities as reviewed by the safety monitoring committee. Secondary end points include a PK study of rhIL7 as well as immunologic studies throughout the duration of the study to assess evidence of IL7 biologic activity with markers of T cell activation, proliferation and differentiation as well as expression of the alpha chain of the IL7 receptor.

This is an Adult AIDS Clinical Trial Group (AACTG) study and the NIAID will participate as a site. The NIAID site will follow all NIAID IRB reporting requirements and all grade 1 and 2 toxicities will be included in the annual review. Children will be excluded and a separate study will be required in the future after the safety and biologic activity of this agent is established in adults.

The study will enroll a total of 40-80 patients followed for a total of eight weeks, with approximately 15-20 anticipated to enroll in our site.

ELIGIBILITY:
INCLUSION CRITERIA:

HIV-1 infection, as documented by any licensed ELISA test kit, and confirmed by Western blot at any time prior to study entry.

Current treatment with potent ART, defined as any protease inhibitor (PI)-based or non-nucleoside reverse transcriptase inhibitor (NNRTI)-based regimen consisting of at least three antiretroviral drugs, for at least 12 months prior to study entry and stable (i.e., no change in dose) for at least 3 months prior to study entry.

Note: Changes in a prior potent ART for purposes of simplification to a two-drug regimen that includes a ritonavir (RTV)-boosted PI and efavirenz will be allowed. RTV-boosted PIs will be considered one antiretroviral drug.

Screening CD4+ cell count greater than or equal to 100 cells/mm(3) obtained within 3-42 days prior to study entry at any CLIA-certified or equivalent laboratory.

Screening HIV-1 RNA less than or equal to 50,000 copies/mL obtained within 3-42 days prior to study entry using an ultrasensitive assay at any CLIA-certified or equivalent laboratory.

Note: If HIV-1 RNA is greater than 400 copies/mL, an ultrasensitive assay is not required at screening.

Documentation that the pre-entry HIV-1 RNA blood draw was obtained within 2-14 days prior to study entry at any CLIA-certified or equivalent laboratory.

Documentation that the pre-entry CD4+/CD8+ blood draw was obtained within 2-14 days prior to study entry at any CLIA-certified or equivalent laboratory.

Laboratory values obtained within 3-42 days prior to study entry:

Absolute neutrophil count (ANC) greater than or equal to 1500/mm(3).

Hemoglobin greater than or equal to 10.0 g/dL.

Platelet count greater than or equal to 100,000/mm(3).

Creatinine less than or equal to 1.5 x upper limit of normal (ULN).

AST (SGOT), ALT (SGPT), and alkaline phosphatase less than or equal to 2 x ULN.

Total bilirubin less than or equal to 2.0 x ULN.

Serum lipase less than or equal to 1.5 x ULN.

Prothrombin time and partial thromboplastin time (PT/PTTT) less than 1.5 x ULN.

Note: For subjects receiving atazanavir or indinavir, total bilirubin less than or equal to 4.0 x ULN.

Female study subjects of reproductive potential (defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months or have not undergone a sterilization procedure (hysterectomy or bilateral oophorectomy), must have a negative serum or urine pregnancy test within 3-42 days prior to study entry.

All study subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, or in vitro fertilization).

If participating in sexual activity that could lead to pregnancy, the study subject must agree that two reliable methods of contraception will be used simultaneously while receiving the protocol-specified medication(s) and for 8 weeks after stopping the medication(s):

Condoms (male or female) with or without a spermicidal agent. Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission.

Diaphragm or cervical cap with spermicide.

IUD.

Hormonal-based contraceptive.

Study subjects who are not of reproductive potential (girls who have not reached menarche, women who have been post-menopausal for at least 24 consecutive months, women who have undergone hysterectomy or bilateral oophorectomy, or prepubescent boys or men who have documented azoospermia) are eligible without requiring the use of contraceptives. Written or oral documentation communicated by clinician or clinician's staff of one of the following:

Physician report/letter.

Operative report or other source documentation in the subject's record (a laboratory report of azoospermia is required to document successful vasectomy).

Discharge summary.

Laboratory report of azoospermia.

FSH measurement elevated into the menopausal range as established by the reporting laboratory.

Karnofsky performance score greater than or equal to 80 obtained within 3-42 days prior to study entry.

Men and women age greater than or equal to 18 years.

Ability and willingness of subject or legal guardian/representative to give written informed consent.

EXCLUSION CRITERIA:

Any history of AIDS-defining illnesses (Category C) during the 12 months prior to study entry. Category C includes the following conditions:

Candidiasis of bronchi, trachea, or lungs;

Candidiasis, esophageal;

Cervical cancer, invasive;

Coccidioidomycosis, disseminated, or extrapulmonary;

Cryptococcosis, extrapulmonary;

Cryptosporidiosis, chronic intestinal (greater than 1 month's duration);

Cytomegalovirus disease (other than live, spleen, or nodes);

Cytomegalovirus retinitis (with loss of vision);

Encephalopathy, HIV-related;

Herpes simplex: chronic ulcer(s) (greater than 1 month's duration); or bronchitis, pneumonitis, or esophagitis;

Histoplasmosis, disseminated, or extrapulmonary;

Isosporiasis, chronic intestinal (greater than 1 month's duration);

Kaposi's sarcoma;

Lymphoma, Burkitt's (or equivalent term);

Lymphoma, immunoblastic (or equivalent term);

Lymphoma, primary, of brain;

Mycobacterium avium complex or M. Kansasii, disseminated, or extrapulmonary;

M. tuberculosis, any site (pulmonary or extrapulmonary);

Mycobacterium, other species, or unidentified species, disseminated, or extrapulmonary;

Pneumocystis carinii pneumonia;

Pneumonia, recurrent;

Progressive multifocal leukoencephalopathy;

Salmonella septicemia, recurrent;

Toxoplasmosis of brain;

Wasting syndrome due to HIV.

Note: Subjects whose sole AIDS-defining illness is Kaposi's sarcoma limited to the skin and who are not anticipated to require systemic chemotherapy may be allowed into the study after discussion with the protocol chairs. Eligible subjects with a history of any AIDS-defining illness (Category C) (greater than 12 months prior to study entry) will be allowed to enroll as long as their screening CD4+ cell count is greater than or equal to 200 copies/mm(3) and was performed at any CLIA-certified or equivalent laboratory.

Palpable lymphadenopathy greater than 2.0 cm.

Breast-feeding.

Known allergy/sensitivity to study drug or its formulations.

Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.

Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 28 days prior to study entry.

Use of any interleukins at any time prior to study entry.

Use of systemic cancer chemotherapy, systemic investigational agents, or immunomodulators (growth factors, systemic corticosteroids, HIV vaccines, immune globulin, and interferons) within 90 days prior to study entry.

Use of heparin within 96 hours prior to study entry or the anticipated need to use heparin within the 96 hours after rhIL-7/placebo injection.

History of malignancy (except basal carcinoma of the skin or Kaposi's sarcoma) including any history of hematologic malignancies and lymphomas.

Splenomegaly (defined as spleen with cephalocaudad diameter greater than 14 cm on ultrasound) and/or proliferative hematologic diseases.

History of hypercoagulability (deep vein thrombosis or pulmonary embolism).

History of seizure disorder.

History of extensive psoriasis, Crohn's disease, uveitis, or other autoimmune disease having induced severe complications.

Significant psychiatric, cardiac, pulmonary, thyroid, renal, or neurological (peripheral or central) disease requiring therapy or severe disorders of hemostasis.

A resting systolic blood pressure greater than 140 or a resting diastolic blood pressure greater than 90.

Note: Blood pressure level must be in the presence of standard anti-hypertensive therapy OR the absence of any anti-hypertensive therapy.

Positive hepatitis B surface antigen or positive hepatitis C antibody at screening.

Plan to start new ART within 8 weeks after study entry.

Lack of adequate venous access and/or inadequate subcutaneous fat tissue that, in the opinion of the investigator, would interfere with study requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2005-03; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Komschlies KL, Grzegorzewski KJ, Wiltrout RH. Diverse immunological and hematological effects of interleukin 7: implications for clinical application. J Leukoc Biol. 1995 Dec;58(6):623-33. doi: 10.1002/jlb.58.6.623. PMID 7499959
- [Background] Benjamin D, Sharma V, Knobloch TJ, Armitage RJ, Dayton MA, Goodwin RG. B cell IL-7. Human B cell lines constitutively secrete IL-7 and express IL-7 receptors. J Immunol. 1994 May 15;152(10):4749-57. PMID 8176200
- [Background] Pandey A, Ozaki K, Baumann H, Levin SD, Puel A, Farr AG, Ziegler SF, Leonard WJ, Lodish HF. Cloning of a receptor subunit required for signaling by thymic stromal lymphopoietin. Nat Immunol. 2000 Jul;1(1):59-64. doi: 10.1038/76923. PMID 10881176